CLINICAL TRIAL: NCT06818994
Title: Safety and Efficacy of Psilocybin-assisted Psychotherapy for Demoralization Syndrome in Patients Diagnosed With Advanced Stage Cancer: a Pilot Study
Brief Title: Safety and Efficacy of Psilocybin-assisted Psychotherapy for Demoralization Syndrome in Patients Diagnosed With Advanced Stage Cancer
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Gustavo Vazquez (Other)
Responsible Party: Sponsor-Investigator, Gustavo Vazquez, Professor of psychiatry at Queen's University, Queen's University
Organization: Queen's University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 65563
Record Dates: First submitted 2025-02-05; First posted 2025-02-11 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-01

CONDITIONS: Demoralization; Safety

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- advanced cancer participants (Experimental)
  Interventions: Drug: Psilocybin-assisted Psychotherapy

INTERVENTIONS:
Drug: Psilocybin-assisted Psychotherapy — The intervention will be psilocybin-assisted psychotherapy. The first treatment period will include four preparation sessions with Managing Cancer and Living Meaningfully (CALM) therapy elements. The psilocybin dosing session will take place after these preparation sessions are completed. The dosing session will include an in-person visit lasting approximately 8 hours in which the participant will receive a capsule of psilocybin 25 mg under constant supervision of therapists. The following day, the first integration session will take place and two weeks later the second integration session along with CALM will be conducted. Participants who show a partial response will be offered a second dosing session, entering the second treatment period. The second treatment period includes a second dosing session using the same dose and safety measures as the first one. It will also be followed by an integration session the following day, and a second integration session with CALM two weeks later.

SUMMARY:
Demoralization syndrome is frequently present in palliative care and oncology patients. In particular, up to a third of patients diagnosed with cancer will experience demoralization due to their illness. The relevance of demoralization syndrome in oncology is tied to this syndrome's association with other mental health ailments such as depression, anxiety, suicidal ideation, and quality of life. Unfortunately, so far no pharmacological strategy has been devised for demoralization, and only a few psychotherapeutic approaches have been trialed in this population, though no psychotherapeutic treatments have been tested for demoralization specifically. The new wave of psychedelic research has been showing encouraging results in a broad spectrum of psychiatric diagnosis, including depression and anxiety in patients diagnosed with cancer and other life-threatening diseases. To date, no clinical trials have been published in which the potential therapeutic effects of psychedelics are explored for the treatment of demoralization syndrome. The aim of this open label pilot study is to assess the safety and efficacy of psilocybin-assisted psychotherapy as a treatment for demoralization syndrome in patients diagnosed with cancer. Fifteen participants between the ages of 18 to 70 years with advanced stage cancer and demoralization syndrome will be enrolled in a treatment program which will include 6 psychotherapeutic sessions and one psilocybin (25 mg) dosing session. Our outcome of interest will be a decrease in demoralization, as measured by the Demoralization Scale at baseline and at the end of the study, and adverse events registration. Other measures of interest include Hamilton Depression Rating Scale, Hamilton Anxiety Rating Scale, and the Columbia Suicide Severity Rating Scale. Those patients with partial response a month after the psilocybin intervention will be offered the possibility of a second psilocybin 25 mg dosing session.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with advanced stage cancer (stages 3 and 4)
* Aged between 18 and 70 years.
* Moderate-to-severe demoralization as measured by Demoralization Scale≥ 30
* English proficiency
* Ability to understand and the willingness to sign a written informed consent document.
* Individuals of child-bearing potential who are sexually active must agree to use an acceptable contraceptive method (hormonal or barrier method of birth control; abstinence) throughout their participation in the study. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled in this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of psilocybin administration.

Exclusion Criteria:

* Condition impairing oral intake or digestive absorption.
* Primary brain tumor.
* Presence of delirium.
* Significant suicide risk as defined by suicidal ideation with intent and a plan.
* Current or past history of schizophrenia, psychotic disorder, bipolar disorder, delusional disorder, paranoid personality disorder, schizoaffective disorder, or borderline personality disorder, as assessed by medical history.
* Patients with first-degree relatives with schizophrenia or bipolar disorder
* Previous diagnosis of epilepsy, stroke or Transient Ischemic Attack (TIA), dementia, and Parkinson's disease.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to psilocybin.
* Other personal circumstances and behavior that would limit compliance with study requirements or that are judged by the study psychiatrist and/or principal investigator to be incompatible with establishing rapport or safe exposure to psilocybin.
* Potential for adverse drug-drug interactions. Concomitant medications with significant potential to interact with study medications will be exclusionary if they cannot be tapered. These include the following:

  * MAO inhibitors
  * Patients currently on antipsychotics (e.g. first and second generation) when taken regularly (6 weeks or less prior to screening visit)
  * Mood stabilizers (e.g. lithium, valproic acid, lamotrigine)
  * Aldehyde dehydrogenase inhibitors (e.g. disulfiram)
  * Significant inhibitors of UGT 1A0 or UGT 1A10
* Patients who have elevated AST and ALT five times above the normal laboratory limit on their last available bloodwork performed at screening and patients with symptoms suggestive of liver failure including confusion, asterixis or jaundice.
* Any other clinically significant cardiovascular, pulmonary, gastrointestinal, hepatic, renal condition or any other unstable condition that, in the opinion of the principal investigator, may interfere with the interpretation of the study results or constitute a health risk for the participant if he/she takes part in the study. This may include but is not limited to clinical symptoms or recent history of significant tachyarrhythmias; severe angina or myocardial ischemia; poorly controlled congestive heart failure; poorly controlled hypertension; poorly controlled hypo- or hyperthyroidism; uncontrolled diabetes; severe renal or liver dysfunction; acute respiratory failure; sepsis; history of cerebral aneurysms; glaucoma; increased intracranial pressure and any intracranial mass.
* Women who are pregnant, nursing, or planning a pregnancy.
* Use of a classic psychedelic or MDMA in the last 12 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Demoralization Scale | From enrollment to the end of the follow up period at week 16 or 19
  Demoralization Scale is a 24-item Likert scale. Items are scored on a 5-point scale from 0 (never) to 4 (all the time), in which higher scores are associated with higher demoralization. Scores can range from 0 to 96. A cut-off point of ≥ 30 in this scale is considered as high demoralization and will be used for participant inclusion in the study.
Adverse Events (AEs) and Serious Adverse Events (SAEs) register | From enrollment to the end of the follow up period at week 16 or 19

SECONDARY OUTCOMES:
Hamilton Anxiety Rating Scale | From enrollment to the end of the follow up period at week 16 or 19
  The Hamilton Anxiety Rating Scale is a 14-item Likert scale. Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56. Higher scores are associated with increased symptom severity, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
Hamilton Depression Rating Scale | From enrollment to the end of the follow up period at week 16 or 19
  The Hamilton Depression Rating Scale is a 17-item Likert scale. Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-68. Higher scores are associated with increased symptom severity.
Columbia Suicide Severity Rating Scale | From enrollment to the end of the follow up period at week 16 or 19
  Columbia Suicide Severity Rating Scale includes ten categories, all of which maintain binary responses (yes/no) to indicate a presence or absence of suicidal behavior. Affirmative answers are associated with higher suicidality

CONTACTS AND LOCATIONS:
Locations (1):
- Queen's University, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No